CLINICAL TRIAL: NCT04488458
Title: Treatment of Periprosthetic Joint Infections Guided by Minimum Biofilm Eradication Concentration (MBEC) in Addition to Minimum Inhibitory Concentration (MIC); a Prospective Randomized Clinical Trial
Brief Title: Susceptibility Testing of Biofilm to Guide Treatment of Periprosthetic Joint Infections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-01471
Record Dates: First submitted 2020-07-10; First posted 2020-07-28 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-07

CONDITIONS: Prosthetic Joint Infection; Prosthetic Infection; Hip Prosthesis Infection; Knee Prosthesis Infection
Keywords: staphylococci; biofilm; antimicrobial resistance; periprosthetic infection
MeSH Terms: interventions — Microbial Sensitivity Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBEC and MIC susceptibility testing (Experimental): For all administered antimicrobials staphylococcal strains must be susceptible in disc diffusion tests/MIC, regardless of MBEC-level. Antibiotic combinations will be selected from 5 already recommended non-cell wall active anti-staphylococcal antibiotics with high per-oral bio-availabilities and acceptable bone penetration used in the treatment of PJIs: rifampicin, fusidic acid, ciprofloxacin/levofloxacin and clindamycin.
  MBEC cut-off for replacement with 2nd or 3rd line antibiotic: RIF MBEC/MIC > 8; LEV MBEC/MIC > 5; FUS MBEC/MIC > 3; CLI MBEC/MIC > 4; LIN MBEC/MIC > 2; T/S MBEC > MIC
  Second line of treatment:
  RIF and Fusidic acid 500 mg TID (ter in die) RIF and Clindamycin 450 - 600 mg TID LEV and Fusidic acid 500 mg TID LEV and Clindamycin 450 mg TID
  Third line of treatment:
  Linezolid 600 mg BID (bis in die) Sulfamethoxazole/Trimethoprim 800/160 mg TID Clindamycin 450 mg TID and Fusidic acid 500 mg TID
  Interventions: Diagnostic Test: MIC or MBEC+MIC based treatment algorithm
- MIC susceptibility testing (Active Comparator): If the causative bacterium is susceptible according to MIC diagnostics, the patient will follow the first line of treatment: Rifampicin 750-900 mg/day + Levofloxacin 750 mg BID
  Interventions: Diagnostic Test: MIC or MBEC+MIC based treatment algorithm

INTERVENTIONS:
Diagnostic Test: MIC or MBEC+MIC based treatment algorithm — i) Non cell wall active standard of care antibiotic combination (MIC-guided) for 6 weeks.
  ii) Non cell wall active antibiotic combination according to a MBEC-based decision algorithm for 6 weeks.

SUMMARY:
The overall purpose of this clinical treatment research project is to explore novel diagnostics that can guide the treatment of infections associated to orthopaedic implants, in order to improve patient outcomes and reduce the development of antibiotic resistance.

The project aims are:

(i) To improve the current diagnostic approaches and treatments of periprosthetic joint infections (PJI) (ii) To investigate the pathogenesis of PJI through the characterization of the virulence carried by the causative pathogens

This multidisciplinary project addresses implant-associated infection and its contribution to increasing antibiotic resistance. Both lead to longer hospital stays, higher medical costs and increased morbidity and mortality. Antibiotic resistance is globally considered as one of the greatest and most urgent risk in medicine. Implant-associated infections are commonly caused by biofilms. Biofilms can be described as 'a community of bacterial cells connected by their secreted extracellular matrix'. Since antibiotics are designed to fight planktonic free-living bacteria, studying antibiotic resistance in biofilm communities poses a paradigm shift. Furthermore, bacteria in biofilms are up to 1000 times more resistant to antibiotics than planktonic bacteria. Mechanisms involved in a biofilm infection also play a crucial role in the development of antibiotic resistance. Hospital-acquired infections are the fourth leading cause of disease and 70% are associated with medical implants and caused by staphylococcal biofilms. In addition, the level of antimicrobial resistance in bacteria causing implant-associated infections has increased worldwide, leaving patients with fewer treatment options.

In this study the investigators will randomize patients with PJI to either standard MIC susceptibility or MIC and MBEC susceptibility guided treatment with oral antibiotic combinations; (i) Non cell wall active standard of care antibiotic combination (MIC-guided) for 6 weeks.

(ii) Or; non cell wall active antibiotic combination according to a MBEC-based decision algorithm for 6 weeks.

In this pilot project, the primary endpoint is how often treatment changes with the MBEC susceptibility testing compared to only MIC-susceptibility testing.

DETAILED DESCRIPTION:
In the infectious process, biofilms may form early on biomaterials. There is ample evidence to the several-fold increase in antimicrobial concentrations required to eradicate even immature biofilms. In clinical practice the choice of antimicrobials is guided by susceptibility testing based on minimum inhibitory concentrations (MIC), which poorly reflect the increased antimicrobial resistance in biofilms. Minimum biofilm eradicating concentrations (MBEC) might better correspond to in vivo efficacy in the treatment of PJI, and other biofilm-centred infections. There is a need to develop methods, which are reproducible, low-cost, and time-efficient, for in vitro susceptibility testing of clinical biofilm bacteria.

This prospective randomized study aim to compare antibiotic treatment regimens for PJI guided by MIC or MBEC combined with MIC, and how it affects infection resolution, drug tolerability and relapse strain resistance patterns.

The investigors hypothesize that a standardised surgical debridement, antibiotics and implant retention (DAIR) for PJI followed by antibiotic guiding MBEC-diagnostics on deep tissue specimens will increase treatment efficacy and decrease the incidence of infection relapses compared to standard of care.

Following standardised debridement and 14 days of parenteral antibiotics; cloxacillin for methicillin sensitive staphylococci or vancomycin for methicillin resistant staphylococci, patients will be randomized to receive oral antibiotic combinations with either cell wall active standard of care antibiotic combination (MIC-guided) for 6 weeks or non cell wall active antibiotic combination according to a MIC- and MBEC-guided decision algorithm for 6 weeks.

Patients will be included at the Orthopaedic Infection Centre (OIC), Sahlgrenska University Hospital/Mölndal, which is a unit dedicated to optimizing management of orthopaedic infections. Patient consent acquisitions and randomisations (20 patients in each group) will be performed during post-operative hospitalisation. MIC determination and disk diffusion will be performed at the SWEDAC (Swedish Accreditation Body) certified clinical bacteriological laboratory. At the department of Biomaterials (University of Gothenburg), a previously developed clinical diagnostic tool will be employed for the MBEC determination. It consists of the combination of the Calgary Biofilm Device (MBECTM P&G Assay, Innovotech) and a custom-made susceptibility plate (Substrata department, Sahlgrenska Hospital) with 6 antimicrobial agents commonly used to treat orthopaedic infections.

Inclusion and exclusion criteria are described in section "Eligibility".

The primary and secondary endpoints are described in section "Outcome measures".

Treatment criteria: for all administered antimicrobials staphylococcal strains must be susceptible in disc diffusion tests/MIC, regardless of MBEC-level. Antibiotic combinations will be selected from 5 already recommended non-cell wall active anti-staphylococcal antibiotics with high per-oral bio-availabilities and acceptable bone penetration used in the treatment of PJIs: rifampicin (RIF), fusidic acid (FUS), ciprofloxacin (CIP)/levofloxacin (LEV) and clindamycin (CLI).

Clinical breakpoints are expressed as MIC (EUCAST and CLSI) but are based on more than MIC distributions (epidemiological cut-off) namely:

* Pharmacokinetic and pharmacodynamic analyses of the antibiotic.
* Relation between MIC and probability of cure in clinical trials.

If likely effective according to EUCAST clinical breakpoints, antibiotics are further ranked in the MBEC treatment algorithm by bone penetration/susceptibility range and semi-arbitrarily by clinical efficacy in prosthetic joint infections.

MBEC/MIC cut-off for replacing Rifampicin despite susceptibility according to MIC:

* C-Max (oral dose of 750 mg) 10 mg/L x 0.4 (Bone/Serum) = 4 mg/L
* RIF-MIC clinical breakpoint for staphylococci is 0.5 mg/L.
* Clinical efficacy factor 1.
* MBEC/MIC ≥ 8 times MIC.

MBEC/MIC cut-off for replacing Levofloxacin despite susceptibility according to MIC:

* C-Max (oral dose of 750 mg) 12 mg/L x 0.6 (Bone/Serum) = 7,2 mg/L
* LEV-MIC breakpoint for staphylococci is 1 mg/L
* Clinical efficacy factor 0,75.
* MBEC/MIC ≥ 5 x MIC.

MBEC/MIC cut-off for not choosing Fusidic acid as companion drug:

* C-Max (500 mg) 30 mg/L x 0,2 (Bone/Serum) = 6 mg/L
* FUS-MIC breakpoint for staphylococci is 1 mg/L.
* Clinical efficacy factor 0,5.
* MBEC 3 times the MIC or more if better companion drug.

MBEC/MIC cut-off for not choosing Clindamycin as companion drug:

* C-Max (600 mg) 12 mg/L x 0.3 (Bone/Serum) = 3,6 mg/L
* CLI-MIC breakpoint for staphylococci is 0.5 mg/L
* Clinical efficacy factor 0,5.
* MBEC/MIC 4 x MIC or more if better companion drug.

MBEC/MIC cut-off for not choosing Linezolid (LIN) as sole drug:

* C-Max 21 mg/L x 0.4 (Bone/Serum) = 8,4 mg/L
* LIN-MIC breakpoint for staphylococci is 4 mg/L
* Clinical efficacy factor 0,5.
* MBEC 2 times the MIC or more.

MBEC cut-off for not choosing Sulfamethoxazole (SMX)/Trimethoprim (TMP) as sole drug:

* C-Max (3200/640 mg SMX/TMP) is 145 and 7.5 mg/L resp. x 0.25 (Bone/Serum) = 36 and 1,9 mg/L resp.
* SMX/TMP-MIC breakpoint for staphylococci is 2 mg/L. (By EUCAST expressed as the Trimethoprim konc.)
* Clinical efficacy factor 0,5.
* MBEC > MIC
* *Interpret as better than according to justification above.

All follow-up up to one year will be done according to clinical routines.

ELIGIBILITY:
Inclusion Criteria:

* first PJI in hip or knee according to Musculoskeletal Infection Society (MSIS) definitions
* first DAIR
* mono-microbial staphylococcal infection
* 14 days of intravenous treatment with either cloxacillin or vancomycin
* standardized administration of local antibiotics

Exclusion Criteria:

* allergy/previous toxic event/unacceptable drug interaction to most effective antibiotic combination according to either MIC or MBEC
* severe drug interactions to MBEC-guided compound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of changes in antimicrobial regimen other than standard of care | 6 weeks
  Proportions of antimicrobial regimens other than standard of care through application of proposed MBEC-algorithm.

SECONDARY OUTCOMES:
Repeat procedure, relapse or reinfection | 12 months
  Number of repeat procedures, relapses or reinfections, according to MSIS-criteria of PJI
Oxford Hip Score | 12 months
  Hip specific patient-reported outcome measure
EQ-5D | 12 months
  Generic health status patient-reported outcome measure
Time to revision | 12 months
  A shorter time could potentially indicate that the right decision is taken at an earlier stage
Inpatient care | Up to 12 months
  Resource consumption measure (days).
Outpatient visits | Up to 12 months
  Resource consumption measure, number of visits, type of visits.
Discharge destination | Up to 12 months
  Resource consumption measure. The type of facility a patient is discharged to (rehab facility, nursing home, home, home care).
Heath care costs | Up to 12 months
  Compound measure using data from outcome 6-8 (currency EUR).
Development of additional antimicrobial resistance of the relapse causative strain | 12 months
  At relapse surgery, the causative strain will be isolated by new biopsy cultures. Then the susceptibility of the causative strain will be tested again to evaluate any possible emergence of resistance against the antimicrobials previously used in the study. This will confirm if the given antimicrobial treatment has lead to antimicrobial resistance in a potential relapse strain isolated at a later occasion.

OTHER OUTCOMES:
Correlation between the virulence properties of the causative bacteria and patient outcome (infection resolution versus recurrent infection) | 36 months
  The staphylococcal strains isolated from the patients with PJI will be characterised by phenotypic tests and whole genome sequencing to determine their virulence properties and carriage of genes involved in biofilm formation, antimicrobial resistance and production of toxins. Then the particular virulence of the strains will be correlated to the patients outcome, to be able to assess if more virulence carriage correlates to worse outcome (recurrent infection)

CONTACTS AND LOCATIONS:
Locations (1):
- Ortopedi, Sahlgrenska University Hospital, Mölndal, Sweden

IPD SHARING:
Plan to Share IPD: No
The main results will be presented at an aggregated level. In some cases, individual data may be presented (e.g. characteristics of a bacterial strain in relation to clinical outcome), but this information will be unidentified so that it cannot be deduced to the individual.
  All compiled personal data will be stored on a password-protected hospital server that only the research group has access to. No personal data will be reported in publications.
  The results of the study will be documented according to the study protocol and placed in a journal. Participants will be coded in a document together with the social security numbers.
  Information about the participants, their health and the code key will be collected at the Orthopaedic Clinic where it will be treated confidentially and securely for 10 years. The handling of the participants' information is regulated by the Personal Data Act (SFS 1998: 204).

REFERENCES:
- [Background] Zaborowska M, Tillander J, Branemark R, Hagberg L, Thomsen P, Trobos M. Biofilm formation and antimicrobial susceptibility of staphylococci and enterococci from osteomyelitis associated with percutaneous orthopaedic implants. J Biomed Mater Res B Appl Biomater. 2017 Nov;105(8):2630-2640. doi: 10.1002/jbm.b.33803. Epub 2016 Oct 25. PMID 27779811
- [Derived] Tillander JAN, Rilby K, Svensson Malchau K, Skovbjerg S, Lindberg E, Rolfson O, Trobos M. Treatment of periprosthetic joint infections guided by minimum biofilm eradication concentration (MBEC) in addition to minimum inhibitory concentration (MIC): protocol for a prospective randomised clinical trial. BMJ Open. 2022 Sep 15;12(9):e058168. doi: 10.1136/bmjopen-2021-058168. PMID 36109038